CLINICAL TRIAL: NCT01341197
Title: A Pan-detecting Assay Based on Stool Samples for Taiwanese Population
Brief Title: Fecal Screening Assay for Taiwanese Population
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201101016RC
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Advanced Colorectal Neoplasms; Throat Cancer; Esophageal Cancer; Gastric Cancer; Important Lower and Upper Gastrointestinal Tract Lesions
Keywords: Fecal immunochemical test; Guaiac fecal occult blood test; Helicobacter pylori stool antigen test; Mass screening; Bidirectional endoscopy
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects undergoing bidirectional endoscopy and fecal tests: Subjects participating in the health check-up at National Taiwan University Hospital (Health Management Center)
  Interventions: Other: Fecal immunochemical test, guaiac fecal occult-blood test, and Helicobacter pylori stool antigen test
- Patients with screening detected GI tract cancers: Patients with screening detected GI tract cancer, such as throat cancer, esophageal cancer, gastric cancer and colorectal cancers, from other screening sites in Taiwan and were referred to the National Taiwan University Hospital for confirmatory diagnosis and treatment.
  Interventions: Other: Fecal immunochemical test, guaiac fecal occult-blood test, and Helicobacter pylori stool antigen test

INTERVENTIONS:
Other: Fecal immunochemical test, guaiac fecal occult-blood test, and Helicobacter pylori stool antigen test
  Other Names: Fecal immunochemical test: OC-SENSOR; Eiken Chemical Co., Ltd, Tokyo, Japan; Guaiac fecal occult-blood test: Hemoccult SENSA Single Slides, Beckman Coulter Inc., USA; Helicobacter pylori stool antigen test: Easy One Step Test, Firstep Bioresearch, Inc., Taiwan

SUMMARY:
Fecal occult blood test (FOBT) is a convenient tool for the screening of asymptomatic gastrointestinal (GI) bleeding while 「guaiac-based fecal occult test (G-FOBT) 」 is increasingly replaced by the use of an 「immunochemical-based test (I-FOBT) 」 that reacts with human globin, a protein that is digested by upper GI enzymes and is specific for detecting lower GI bleeding. However, in Taiwan, although the incidence of colorectal cancer is rapidly increasing, Helicobacter pylori-related upper GI pathologies remain highly prevalent, which may imply that mass screening solely based on I-FOBT could be insufficient as significant upper GI pathologies can be missed. Since I-FOBT dose not predict upper GI pathologies, the adjuncts of G-FOBT and H. pylori stool-antigen test (HpSA) may be a potential candidate to realize a pan-detecting assay based on stool samples in a population in which both lower and upper GI lesions are equally prevalent.

DETAILED DESCRIPTION:
Background and objective: Fecal occult blood test (FOBT) is a convenient tool for the screening of asymptomatic gastrointestinal (GI) bleeding while 「guaiac-based fecal occult test (G-FOBT) 」 is increasingly replaced by the use of an 「immunochemical-based test (I-FOBT) 」 that reacts with human globin, a protein that is digested by upper GI enzymes and is specific for detecting lower GI bleeding. However, in Taiwan, although the incidence of colorectal cancer is rapidly increasing, Helicobacter pylori-related upper GI pathologies remain highly prevalent, which may imply that mass screening solely based on I-FOBT could be insufficient as significant upper GI pathologies can be missed. Since I-FOBT dose not predict upper GI pathologies, the adjuncts of G-FOBT and H. pylori stool-antigen test (HpSA) may be a potential candidate to realize a pan-detecting assay based on stool samples in a population in which both lower and upper GI lesions are equally prevalent.

Patients: Our study will enroll consecutive subjects participating in the health check-up at National Taiwan University Hospital (Health Management Center), who will undergo I-FOBT, G-FOBT, HpSA, colonoscopy and EGD. The diagnostic values of three fecal testing, alone or in combination, will be respectively evaluated. knowing that subjects who were detected with gastrointestinal tract cancers might be small based on one screening setting, we also recruited patients who were detected with gastrointestinal tract cancers at other screening sites and were referred to the National Taiwan University Hospital for confirmatory diagnosis and treatment. They were also requested to complete the three fecal tests as well as the bidirectional endoscopies; however, it should be noted that, in this group of patients, those who completed only one of the bidirectional endoscopies were still eligible.

Our primary hypothesis was to test whether a guaiac-based test combined with an immunochemical test could help differentiate occult bleeding in the upper gastrointestinal tract from that in the lower gastrointestinal tract. As such a hypothesis would not be held, we also evaluated an alternative choice based on Helicobacter pylori stool antigen test to catching the upper gastrointestinal tract lesions.

ELIGIBILITY:
Inclusion Criteria:

* subjects who received three fecal tests and receive confirmatory endoscopic diagnosis

Exclusion Criteria:

* subjects who had overt gastrointestinal bleeding (e.g., hematemesis, tarry stool, melena, and hematochezia) that would normally push the patients to seek immediate health care instead of participating in screening programs.
* subjects who do not receive the fecal tests
* subjects who do not receive the confirmatory endoscopic diagnosis
* subjects who had undergone gastrectomy or colectomy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study will enroll consecutive subjects participating in the health check-up at National Taiwan University Hospital (Health Management Center), who will undergo a standard protocol, including I-FOBT, G-FOBT, HpSA, face-to-face interviews, blood chemistries, colonoscopy and EGD. Prior to the examination, a self-administered questionnaire will be used to collect information on participants' demographics, social habits, clinical symptoms, and medical/medication histories. To ensure that our study population was asymptomatic and the bleeders were occult, we excluded those who had overt GI symptoms and overt GI bleeding from analyses. During the same period, patients with screening detected GI tract cancers from other screening sites, such as throat cancer, esophageal cancer, gastric cancer, and colorectal cancers, will also be invited to participated in the study. This enrollment was based on insufficient GI cancer case number in the interim analyses based on a single screening site.
Sampling Method: Probability Sample
Enrollment: 3172 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Important Lower and Upper GI tract Lesions | On the day of receving endoscopy
  We define significant lower GI lesions as mass lesions (carcinoma and advanced adenoma), inflammation (erosive esophagitis, ulcer, and colitis), and vascular disorders (vascular ectasia and varices). Hyperplastic polyps are not considered significant lesions. Important upper GI lesions include cancer, esophageal varix, ulcer at least 0.5 cm in diameter with a perceptible depth, and angiodysplasia. Biopsies will be performed over any suspicious lesions for pathological confirmation. Reflux esophagitis with Los Angeles grade A or B severity is not considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chia Lee, MD.PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Lee YC, Chiu HM, Chiang TH, Yen AM, Chiu SY, Chen SL, Fann JC, Yeh YP, Liao CS, Hu TH, Tu CH, Tseng PH, Chen CC, Chen MJ, Liou JM, Liao WC, Lai YP, Wang CP, Ko JY, Wang HP, Chiang H, Lin JT, Chen HH, Wu MS. Accuracy of faecal occult blood test and Helicobacter pylori stool antigen test for detection of upper gastrointestinal lesions. BMJ Open. 2013 Oct 30;3(10):e003989. doi: 10.1136/bmjopen-2013-003989. PMID 24176798